CLINICAL TRIAL: NCT02705781
Title: Functionality and Accuracy of the smARTrack System in Real-Life ICU Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ART Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EXC_SYT_P001
Record Dates: First submitted 2016-02-09; First posted 2016-03-11 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Aspiration Pneumonia
MeSH Terms: conditions — Pneumonia, Aspiration

ARMS (1):
- General (Experimental): One arm study: smARTrack Feeding Tube System.
  Interventions: Device: smARTrack Feeding Tube System

INTERVENTIONS:
Device: smARTrack Feeding Tube System

SUMMARY:
This study conducted in order to validate the functionality and accuracy of the smARTrack™ System in a real-life ICU setting. The smARTrack™ Feeding Tube System is a novel system with nasogastric tube developed by ART Healthcare Ltd, based on sensor-lined tubes that transmit real-time information to an external console. The smARTrack™ feeding tube is equipped with reflux sensors which alert when gastric contents regurgitating into the esophagus. In addition, the smARTrack™ feeding tube is equipped with sensors designed to provide information about the location of the tube thus assisting in reducing the incident of misplacement during first positioning. The smARTrack™ feeding tube is also automatically and in real-time stops feeding if the feeding tube moves out of position during ongoing use or detect gastric content in esophagus. Furthermore, smARTrack™ Feeding Tube System can guide operator to correctly re-position the tube.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years or older
* Patient has already been admitted to ICU
* Patient requires enteral feeding
* Patients receiving PPI therapy
* Informed consent by independent physician and next of kin
* ICU ventilated patients

Exclusion Criteria:

* Patients with anomalies or diseases of the nose, throat, or esophagus and or stomach.
* Patients with known sensitivities or allergies to any of the feeding tube materials
* Inability to place patient is semi-Fowler's position.
* Any clinically significant abnormality upon physical examination which may, in the opinion of the investigator, pose difficulty in inserting the feeding tube (e.g. cervical spine disorder)
* Pregnancy
* Recent abdominal surgery (less than 30 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
System accurately guides correct initial placement | 24-72 hours
  The system is able to accurately guide the user to ensure correct initial placement (verified by X-ray)
System accurately detects tube movement/displacement during ongoing use | 24-72 hours
  The system is able to detect tube movement/displacement during ongoing use (verified by markings on the tube)
System automatically stops feeding when displacement is detected | 24-72 hours
  The system automatically stops feeding when tube displacement is detected
System is able to detect overfeeding | 24-72 hours
  The system is able to detect overfeeding
Occurrence of device related Adverse Events (Safety) | 24-72 hours
  Occurrence of device related adverse events

SECONDARY OUTCOMES:
The system user interface is easy for use | 24-72 hours
  Ease of use of the system and the user interface by subjective questionnaire of staff
Correlation of impedance detected to patient positioning | 24-72 hours
  Recording of impedance detected by the system and correlation to patient positioning
Quantification of the amount of discarded nutritional supplement by implementing GRV test | 24-72 hours
  Quantification of the amount of discarded nutritional supplement by implementing GRV test as needed and according to hospital procedures
Aspiration of gastric contents percentage compared to standard feeding (as reported in literature) | 24-72 hours
  Reduction of aspiration of gastric contents percentage compared to standard feeding (as reported in literature).
Correlation between patient clinical information and the occurrence of reflux and sensors data | 24-72 hours
  Correlation between patient clinical information and the occurrence of reflux and sensors data.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel